CLINICAL TRIAL: NCT05607888
Title: Prospective Observational Study of Sinonasal and Skull-base Tumours Management in a Tertiary Referral Otorhinolaryngology Service
Brief Title: Prospective Study of Sinonasal and Skull-base Tumours Management
Acronym: Sinonasal_Tu
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Domen Vozel, MD, PhD, Domen Vozel, MD, PhD, principal investigator, University Medical Centre Ljubljana
Other Study IDs: Sinonasal tumours
Record Dates: First submitted 2022-10-30; First posted 2022-11-07 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Nasal Neoplasm; Nasal Neoplasm Benign; Skull Base Neoplasms; Skull Base Osteomyelitis; Sinonasal Disorder; Sinus Disease
MeSH Terms: conditions — Nose Neoplasms; Skull Base Neoplasms; Paranasal Sinus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational prospective clinical study aims to describe the epidemiology, management and outcome of patients with sinonasal and skull-base pathology (tumours and diseases with malignant clinical characteristics) in a tertiary otorhinolaryngology referral centre. The main questions it aims to answer are:

* what is the caseload of patients with the included pathology in our centre
* what are the results of management of these cases
* what are the epidemiological characteristics of included patients
* what is the quality of life of included patients.

DETAILED DESCRIPTION:
Sinonasal tumours and tumours that involve the adjacent skull base are rare entities. However, their management necessitates a special knowledge of ENT areas and specifics of sinonasal anatomy and skull base. Due to the heterogeneity of pathological diagnoses of sinonasal and skull-base tumours, one of the main aims of this study is to provide epidemiological characteristics in our geographical area. Furthermore, to compare with other tertiary referral centres, we will analyse management results, which could improve the management of these diseases. Since the sinonasal area and skull base house several important neuroanatomical structures and senses, we aim to provide an analysis of the patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* sinonasal and/or skull-base cancer
* sinonasal disease expanding through the skull-base
* the patient's written informed consent

Exclusion Criteria:

* lateral skull-base disease primarily originating in the temporal bone and without central skull-base involvement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from patients referred to the tertiary otorhinolaryngology referral centre. The referral applies to the in-hospital or outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Absence of the disease | twelve months after the treatment completion
  Absence of the disease after the treatment has been completed
Overall survival | twelve months after the treatment completion
  Survival after the treatment has been completed

CONTACTS AND LOCATIONS:
Overall Officials: Domen Vozel, MD, PhD, Study Director — University Medical Centre Ljubljana; Jure Urbančič, MD, Study Director — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia